CLINICAL TRIAL: NCT01309451
Title: A Single Masked, Randomized Controlled Study to Assess Efficacy of Ozurdex as Adjunct to Avastin Compared With Avastin Alone in the Treatment of Patients With Diabetic Macular Edema
Brief Title: Ozurdex as Adjunct to Avastin Compared to Avastin Alone in Treatment of Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maturi, Raj K., M.D., P.C. (Individual)
Responsible Party: Principal Investigator, Raj K. Maturi, MD, PI, Maturi, Raj K., M.D., P.C.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OA002
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; DME
MeSH Terms: interventions — Bevacizumab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab alone (Active Comparator)
  Interventions: Drug: Bevacizumab
- Combined group (Active Comparator): Bevacizumab plus Ozurdex
  Interventions: Drug: Bevacizumab; Drug: dexamethasone intravitreal implant

INTERVENTIONS:
Drug: Bevacizumab — intravitreal, 1.25mg., monthly
  Other Names: Avastin
Drug: dexamethasone intravitreal implant — 0.7mg, intravitreal every 4 months
  Other Names: Ozurdex
  Arms: Combined group

SUMMARY:
The investigators hypothesize that a combination treatment with Avastin and Ozurdex will result in a more rapid improvement of visual acuity compared to the use of Avastin alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 years or older
* Type 1 or type 2 diabetes
* BCVA score of >24 and <78 letters
* Presence of DME defined as Optical Coherence Tomography Center Subfield Thickness (OCT CST) >250microns

Exclusion Criteria:

* Anti-VEGF intravitreal treatment in last 4 weeks
* Intravitreal steroid treatment in the last 8 weeks
* PRP or Focal laser in last 4 months
* Active iris neovascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Maturi, MD, Principal Investigator — Midwest Eye Institute
Locations (1):
- Raj K. Maturi, MD, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center. The sample size was 40 eyes (30 subjects, 10 subjects had both eyes in study)
Pre-assignment Details: Subjects were randomly assigned to either bevacizumab alone or bevacizumab plus Ozurdex in a 1:1 ratio. When both eyes were eligible, the right eye was randomized and the left eye was assigned to the other group. We had a total of 30 subjects, 10 with both eyes. 19 eyes were in the Bevacizumab Alone group and 21 eyes were in the Combined Group.
Groups:
- Bevacizumab Alone: monthly injection of bevacizumab intravitreally when retreatment criteria met
- Combined Group: bevacizumab plus Ozurdex group received bevacizumab at baseline followed by Ozurdex at the one month visit. Retreatment with bevaciumab given at monthly intervals when retreatment criteria met except for months 5 and 10 when retreatment with Ozurdex was given.
Period: Overall Study
Arm/Group | Bevacizumab Alone | Combined Group
Started | 19 (unit of measure is number of eyes) | 21 (unit of measure is number of eyes)
Completed | 17 (unit of measure is number of eyes) | 18 (unit of measure is number of eyes)
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: The unit of "eyes" is used to described the number of participants since some subjects had both eyes in the study and it is not feasible to separate those into their own group.
Groups:
- Bevacizumab Alone: Bevacizumab only
- Combine Group: Bevacizumab plus Ozurdex
- Total: Total of all reporting groups
Arm/Group | Bevacizumab Alone | Combine Group | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9) | 59 (12) | 60.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: eyes] — The sample size was 40 eyes (30 subjects, 10 subjects had both eyes in study)
  eyes
    United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity (BCVA) Measured Using Early Treatment of Diabetic Retinopathy Study (ETDRS) Methodology at Month 12 Compared to Baseline
Description: Visual Acuity was measured with the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity test. Unit of measure is based on the ETDRS letter score scale, 0-97, where 0 = worst and 97 = best.
Time Frame: baseline to 12 month
Population: The unit of measure is EYES rather than actual number of participants
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Bevacizumab Alone | Combined Group
Number analyzed (Participants) | 19 | 21
letters | 4.9 (12.3) | 5.4 (10.7)

2. Primary Outcome: OCT CST
Description: change in optical coherence tomography central subfield thickness
Time Frame: change in OCT CST from baseline to twelve months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Bevacizumab Alone | Combined Group
Number analyzed (Participants) | 19 | 21
microns | 30 (100) | 45 (107)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Bevacizumab Alone Group: bevacizumab 1.25mg intravitreally
- Combined Group: bevacizumab 1.25mg intravitreally plus Ozurdex THIS GROUP ALSO INCLUDES PARTICIPANTS WHO HAD BOTH EYES IN THE STUDY (they received bevacizumab alone in one eye and bavacizumab + Ozurdex in the other.
Arm/Group | Bevacizumab Alone Group | Combined Group
Serious Adverse Events (participants affected / at risk) | 2/9 | 8/21
Other Adverse Events (participants affected / at risk) | 9/9 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Alone Group (N=9) | Combined Group (N=21)
acute renal insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 1 (1)
cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
generalized weakness (General disorders) | 0 (0) | 1 (1)
worsening of hypertension (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Alone Group (N=9) | Combined Group (N=21)
headaches (Nervous system disorders) | 1 (1) | 1 (1)
renal insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
angina (Cardiac disorders) | 0 (0) | 1 (1)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
blepharitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
osteophyte right foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
canaliculitis (Infections and infestations) | 1 (1) | 0 (0)
carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 2 (2)
congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
contusion left arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
corneal abrasion (Eye disorders) | 1 (1) | 0 (0)
corneal precipatates (Eye disorders) | 0 (0) | 1 (1)
coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
cough (General disorders) | 0 (0) | 2 (2)
cyst lower eyelid (Eye disorders) | 1 (1) | 0 (0)
decreased ability to concentrate (Psychiatric disorders) | 0 (0) | 1 (1)
decreased visual acuity (Eye disorders) | 0 (0) | 1 (1)
degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
dizziness (General disorders) | 2 (2) | 0 (0)
dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
epiretinal membrane (Eye disorders) | 5 (5) | 4 (4)
esophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
esophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
fallen arch left foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
vitreous floater (Eye disorders) | 1 (1) | 4 (4)
peripheral edema (Renal and urinary disorders) | 0 (0) | 1 (1)
fracture ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
suspected glaucoma (Eye disorders) | 1 (1) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
hordeolum lower eyelid (Eye disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
increased intraocular pressure (Eye disorders) | 2 (2) | 6 (8)
infection of toe (Infections and infestations) | 0 (0) | 1 (1)
iritis (Eye disorders) | 0 (0) | 1 (1)
keratitis (Eye disorders) | 0 (0) | 2 (2)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
loss of blood sugar control (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
low back bain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
low tension glaucoma (Eye disorders) | 0 (0) | 1 (1)
macular scar (Eye disorders) | 0 (0) | 1 (1)
magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
nail fungus (Infections and infestations) | 0 (0) | 2 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
neovascularization of retina (Eye disorders) | 3 (3) | 1 (2)
peripheral vascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
poison ivy (Infections and infestations) | 1 (1) | 0 (0)
posterior capsule opacification (Eye disorders) | 0 (0) | 6 (6)
heel discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
laceration right leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
sciatica (Nervous system disorders) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 0 (0) | 5 (5)
sleep apnea (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
ankle sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
subconjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1)
tear film insufficiency (Eye disorders) | 0 (0) | 1 (1)
tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
foot ulcer (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
visual disturbance (Eye disorders) | 1 (1) | 0 (0)
vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1)
worsening of cataract (Eye disorders) | 7 (7) | 8 (8)
worsening of coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
worsening of diabetes mellitus (Endocrine disorders) | 0 (0) | 1 (1)
worsening of hypertension (Cardiac disorders) | 0 (0) | 4 (4)
worsening of peripheral vascular disease (Cardiac disorders) | 0 (0) | 1 (1)
worsening of posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1)
worsening of vitreoretinal traction (Eye disorders) | 0 (0) | 1 (1)
worsening of vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No